CLINICAL TRIAL: NCT04413669
Title: Bronchoscopy Screening of High-risk Population of Lung Cancer With Severe Smoking
Brief Title: Bronchoscopy Screening for High-risk Population of Lung Cancer With Severe Smoking With Negative LDCT Screen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiayuan Sun (Other)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Director, Department of Endoscopy, Shanghai Chest Hospital, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SHCHE201907
Record Dates: First submitted 2020-01-03; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-01

CONDITIONS: Heavy Smoking
Keywords: Heavy smoking; People at high risk for lung cancer; autofluorescence bronchoscopy，AFB; white light bronchoscopy, WLB

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- white light bronchoscopy and autofluorescence bronchoscopy (Experimental): White light bronchoscopy and autofluorescence bronchoscopy were carried out for people at high risk for lung cancer with heavy smoking (smoking history> 400 years).Biopsy was taken for abnormal bronchial mucosa.
  Interventions: Procedure: white light bronchoscopy & autofluorescence bronchoscopy

INTERVENTIONS:
Procedure: white light bronchoscopy & autofluorescence bronchoscopy — White light bronchoscopy and autofluorescence bronchoscopy were carried out，and Take a biopsy for abnormal bronchial mucosa

SUMMARY:
Based on the previous work of LDCT screening, in order to improve the screening rate of central lung cancer for LDCT negative and severe smokers, the investigators plan to conduct China's first large-scale fluorescent bronchoscopy screening test.

DETAILED DESCRIPTION:
CT scan is a commonly used method for clinical screening for early lung cancer, but research shows that LDCT scan has a higher detection rate for peripheral lesions (often adenocarcinoma), and a lower detection rate for central lung cancer (mostly squamous cell carcinoma). Fluorescent bronchoscopy uses the principle of differentiating fluorescence in different tissues to distinguish normal parts from diseased parts. It is often used for screening of central early lung cancer.Based on the results of the investigator's previous research, the investigators plan to conduct a second round of community screening-bronchoscopy screening, and perform white light bronchoscopy and autofluorescence bronchoscopy screening for high-risk groups of lung cancer with heavy smoking (≥400 years) and no obvious lung nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-75 years;
2. have a smoking history of ≥20 pack years; if participants quit smoking, it should be <15 years;
3. Chest LDCT examination within one and a half years without obvious abnormalities or calcified nodules or non-calcified nodules and no signs of malignancy

Exclusion Criteria:

1. Non-smokers or mild smokers;
2. There are contraindications to bronchoscopy, such as active hemoptysis, unstable angina pectoris, coagulation dysfunction, anesthesia allergy, etc .;
3. Refusing to sign informed consent;
4. The operator believes that the patient has other conditions that are not suitable for bronchoscopy.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-12-26 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
The effect of AFB and WLB screening （the positive rate of lung cancer）on LDCT screening negative at high risk for lung cancer was analyzed. | one year
  ALB and WLB were screened for LDCT screening for lung cancer negative severe smokers. The effect of AFB and WLB screening on LDCT screening negative lung cancer at high risk was analyzed.

SECONDARY OUTCOMES:
The diagnostic efficacy of WLB and AFB in lung cancer was compared | one year
  The diagnostic efficacy of WLB and AFB in lung cancer was compared by comparing abnormalities under WLB and AFB and histopathology respectively.
The independent risk factors of lung cancer in high-risk groups were Identified. | one year
  Univariate and multivariate Logistic regression analysis was carried out to screen the independent risk factors of lung cancer in high-risk groups.
RGB（red-green-blue） chrominance spatial differences in normal sites, low-grade preinvasive (LGD), high-grade intraepithelial neoplasia, and invasive cancer was analyzed. | one year
  RGB（red-green-blue） chrominance spatial differences of AFB in normal sites, low-grade preinvasive (LGD), high-grade intraepithelial neoplasia, and invasive cancer was analyzed.
Blood was drawn for liquid molecular detection to identify the molecular markers associated with lung cancer. | one year
  Blood was drawn for liquid molecular detection to identify the molecular markers associated with lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No